CLINICAL TRIAL: NCT04288739
Title: Relationship Between Immunophenotyping and X-inactive Specific Transcript (Xist) Gene in Acute Myeloid Leukemia
Brief Title: Immunophenotyping and Xist Gene in AML
Acronym: Xist
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mahmoud Ali Kassem, Assistant lecturer, Assiut University
Other Study IDs: AssiutU-CP-Xist 90
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood or bone marrow aspirate samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia (AML) group: patients who are diagnosed as Acute Myeloid Leukemia (AML) based on peripheral blood, bone marrow, immunophenotyping and who fulfill the WHO 2016 criteria.
  Complete blood count (CBC), bone marrow aspirate, flow cytometric immunophenotyping, cytogenetic analysis and fluorescence in situ hybridization (FISH) for XIST gene will be performed for all AML patients in the study.
  Interventions: Diagnostic Test: flow cytometric immunophenotyping; Genetic: Xist gene by fluorescence insitu hybridization

INTERVENTIONS:
Diagnostic Test: flow cytometric immunophenotyping — Flow cytometric (FCM) immunophenotypic analysis of peripheral blood or bone marrow aspiration samples will be performed using a panel of monoclonal antibodies (HLA DR, CD34, CD117, Cyto MPO, CD13, CD33, CD3, CD4, CD8, CD10, CD19, CD5, CD14, CD64, CD36, CD235a, cyto CD41, cyto CD61).
Genetic: Xist gene by fluorescence insitu hybridization — Fluorescence in situ hybridization (FISH) is a kind of cytogenetic technique that allows the visualization of defined nucleic acid sequences in particular cellular or chromosomal sites by hybridization of complementary fluorescently labeled probe sequences within intact metaphase or interphase cells.
  The fluorescent probes are nucleic acid labeled with fluorescent groups and can bind to specific DNA/RNA sequences. Fluorescence microscopy can be used to find out where the fluorescent probe is bound to the chromosomes.
  Other Names: FISH

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous disorder characterized by clonal expansion of myeloid progenitors (blasts) in the bone marrow and peripheral blood.Several studies have reported correlations of aberrantly expressed markers by flowcytometry with clinical outcome in AML. X-inactive specific transcript RNA was one of the first long noncoding RNAs (lncRNAs) to be discovered in the early 1990s. Xist RNA is the master regulator of XCI, the epigenetic process that equalizes the dosage of X-linked genes between female (XX) and male (XY) mammals. Yildirim et al., (2013) deleted Xist in the blood compartment of mice and demonstrated that mutant females developed a highly aggressive myeloproliferative neoplasm and myelodysplastic syndrome (mixed MPN/MDS) with 100% penetrance.

Their study implies that human hematologic cancers may result from overdosage of X, either from Xist loss on Xi or from duplication of Xa. And they proposed that carcinogenesis is driven by a series of changes occurring in the HSC and further accumulated in mature hematopoietic cells. These changes are initiated by loss of Xist, which leads to progressive X reactivation, which in turn induces a cascade of unfavorable genome-wide changes that include dysregulation of genes involved in DNA replication, chromosome segregation, cell-cycle checkpoints, and hematopoiesis. A failure of HSC maturation and loss of long-term HSC in the marrow progressively shift hematopoiesis to extramedullary sites resulting in extra medullary hematopoiesis (EMH), thereby causally linking the X chromosome to cancer in mice. Thus, they concluded that Xist RNA not only is required to maintain XCI but also suppresses cancer in vivo.

Indeed, the emerging role of aberrant gene dosage in diseases, whether of the X chromosome or for autosomes, brings with it the possible application of drugs that impact on epigenetic regulators in potential therapeutic strategies.

To date, there are no published studies on human about Xist gene and its relationship with the immunophenotyping in AML patients. So, this will be the first study designed to explain its unexplored pathway in AML and detect its prognostic role and immunophenotypic association.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous disorder characterized by clonal expansion of myeloid progenitors (blasts) in the bone marrow and peripheral blood. with high mortality and variable prognosis. AML is the most common acute leukemia in adults, accounting for ~ 80 percent of cases in this group. There are approximately 19,520 new cases of AML in the United States (US) each year and 10,670 deaths from AML. In Egypt, the incidence of AML was 0.96% for males and 1.14% for females according to the results of the National Population-Based Registry Program of Egypt (2008-2011). Diagnosis of AML based on morphological diagnosis with proliferation of blast cells ≥ 20% of marrow cells, flow cytomtric immunophenotyping and cytogenetic abnormalities.

Immunophenotyping via flow cytometry comprises an additional fast technique to predict outcome in AML, although only few markers are yet established as prognostic factors in clinical routine diagnosis, despite the fact that new and rapidly available markers are needed to improve the treatment decisions in AML patients. This is even more since therapy in AML patients must be initiated immediately after diagnosis. AML blasts express antigens found also on healthy immature myeloid cells, including common differentiation (CD) markers CD13, CD33 and CD34. Other cells markers are expressed depending on the morphological subtype of AML and stage of differentiation block such as monocytic differentiation markers (CD4, CD14, CD11b, CD11c, CD64, CD36), erythroid (CD36, CD71) and megakaryocytic markers (CD41a and CD61).

Non-random chromosomal abnormalities (e.g., deletions, translocations) are identified in approximately 52% of all adult primary AML patients and have long been recognized as the genetic events that cause and promote this disease. Certain cytogenetic abnormalities, including the t(8;21)(q22;q22), t(15;17)(q22;q12) and inv(16)(p13.1;q22) are associated with longer remission and survival, while alterations of chromosomes 5, 7, complex karyotype (described as >3 chromosomal abnormalities) and 11q23 are associated with poor response to therapy and shorter overall survival.

Several studies have reported correlations of aberrantly expressed markers with clinical outcome in AML. For example, CD7 and CD25 expression has been associated with poor prognosis in normal karyotype (NK) AML. The IL3 receptor alfa (CD123) is overexpressed in 45% of AML patients, and this higher expression has also been associated with poor outcome and correlated with mutations in the fms-like tyrosine kinase receptor (FLT3) gene. A consistent antigenic profile with high CD33 expression has also been associated with AML with mutated nucleophosmin (NPM1). Lo-Coco et al., (2015) results suggest that the CD34/25/123/99+ve leukemia-associated immunophenotypes (LAIPs) is strictly associated with FLT3-ITD positive cells. This identification through multiparametric flow cytometry at diagnosis of an immunophenotypic fingerprint associated with these subclones is a novel and simplified tool with improved sensitivity to unravel these clones and allowing patient stratification and risk adapted treatment with potential impact on outcome of the disease.

At present, the etiological agent and pathogenesis of AML are not entirely clear, only few AML cases can be accurately classified through traditional cellular morphological classification. Thus, it is very difficult to judge the disease condition and predict prognosis. Improper expression of specific genes is a common finding in AML and may induce clinically relevant biological subsets. Consequently, identification of novel biomarkers which could predict outcome or guide treatment choice will make more contribution to the clinical management of AML.

X chromosome aneuploidies have long been associated with human cancers, but causality has not been established. In mammals, X chromosome inactivation (XCI) is triggered by X-inactive specific transcript (Xist) RNA to equalize gene expression between the sexes. In humans, one X chromosome is inactivated (Xi) in every female cell in order to achieve transcriptional balance. An X-linked inactivation centre (XIC) is responsible for the initiation of X inactivation. The exact size of the XIC is unclear but it includes the Xistgene at Xq13.2. This encodes a large non-coding RNA that is initially expressed on both X chromosomes before ceasing expression on the active X and becoming upregulated on the X that is to become inactivated. The Xist RNA product coats the future Xi chromosome, spreading out from the XIC.

X-inactive specific transcript RNA was one of the first long noncoding RNAs (lncRNAs) to be discovered in the early 1990s, a decade before the Human Genome Project (HGP) revealed that the large majority of our genome accounts for noncoding sequences. Xist is a 19 kb, spliced, untranslated regulatory transcript that coats the X chromosome from which it is expressed in cis. Xist RNA is the master regulator of XCI, the epigenetic process that equalizes the dosage of X-linked genes between female (XX) and male (XY) mammals. Deletion of the Xist gene results in skewed inactivation of the wild type X chromosome, indicating that this locus is essential for gene silencing.

The early transgenic studies also unveiled two key features of Xist's function. First, the ability of Xist RNA to trigger gene silencing is strictly dependent on the developmental context. Second, Xist has different tasks, such as cis-localization to the chromosome from which it is expressed and the ability to trigger gene silencing, and these tasks are mediated by genetically independent domains of the RNA. Moreover, inappropriate silencing of human Xist results in qualitatively aberrant stem cells. Whereas Xist has been investigated extensively in cell culture, in vivo studies have been limited, however, none of these studies has been done in human.

In some cases, Xist RNA mislocalisation and sporadic Xi reactivation has been observed. For example, one study on an ovarian cancer cell line, showed a disruption of Xist expression and potential reactivation of the Membrane Palmitoylated Protein-1 (MPP1) (p55) gene. Previous study showed that the inactive X chromosome is genetically unstable in cancer as this study reporting an higher mutations rate on the inactive X compare to rest of the genome.

Xist deletion in the blood compartment of mice demonstrated that mutant females developed a highly aggressive myeloproliferative neoplasm and myelodysplastic syndrome (mixed MPN/MDS) with 100% penetrance. Significant disease components include primary myelofibrosis, leukemia, histiocytic sarcoma, and vasculitis. They found that proliferative and dysplastic changes were present in all hematopoietic cell types. Also, Xist-deficient hematopoietic stem cells (HSCs) showed aberrant maturation and age-dependent loss of long-term HSCs.

Their study implies that human hematologic cancers may result from overdosage of X, either from Xist loss on Xi or from duplication of Xa. And they proposed that carcinogenesis is driven by a series of changes occurring in the HSC and further accumulated in mature hematopoietic cells. These changes are initiated by loss of Xist, which leads to progressive X reactivation, which in turn induces a cascade of unfavorable genome-wide changes that include dysregulation of genes involved in DNA replication, chromosome segregation, cell-cycle checkpoints, and hematopoiesis. A failure of HSC maturation and loss of long-term HSC in the marrow progressively shift hematopoiesis to extramedullary sites resulting in extra medullary hematopoiesis (EMH), thereby causally linking the X chromosome to cancer in mice. Thus, they concluded that Xist RNA not only is required to maintain XCI but also suppresses cancer in vivo.

Indeed, the emerging role of aberrant gene dosage in diseases, whether of the X chromosome or for autosomes, brings with it the possible application of drugs that impact on epigenetic regulators in potential therapeutic strategies.

To date, there are no published studies on human about Xist gene and its relationship with the immunophenotyping in AML patients. So, this will be the first study designed to explain its unexplored pathway in AML and detect its prognostic role and immunophenotypic association.

ELIGIBILITY:
Inclusion Criteria:

* AML patients, who fulfill the WHO 2016 criteria

Exclusion Criteria:

* patients with other hematological nepolasms (ALL,CLL, plasma cell myeloma)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AML patients, who fulfill the WHO 2016 criteria
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-10-02 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify Xist gene by FISH in AML | 2 years
  Identify X- inactive specific transcript (Xist) gene by fluorescence insitu hybridization (FISH) in AML
Integrating multiple strategies ( immunophenotypic fingerprint by flowcytometry and Xist gene by FISH) in AML | 2 years
  Integrating multiple strategies by Identification through multiparametric flow cytometry atdiagnosis of an immunophenotypic fingerprint associated with Xist gene abnormalities, detected by FISH, as a novel and simplified tool with improved sensitivity, to detect these abnormalities may allowing patient stratification and risk adapted treatment with potential impact on outcome of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban R. Helal, MD, Study Director — faculty of medicine
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Estey EH. Acute myeloid leukemia: 2019 update on risk-stratification and management. Am J Hematol. 2018 Oct;93(10):1267-1291. doi: 10.1002/ajh.25214. PMID 30328165
- [Background] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Background] Cronin KA, Lake AJ, Scott S, Sherman RL, Noone AM, Howlader N, Henley SJ, Anderson RN, Firth AU, Ma J, Kohler BA, Jemal A. Annual Report to the Nation on the Status of Cancer, part I: National cancer statistics. Cancer. 2018 Jul 1;124(13):2785-2800. doi: 10.1002/cncr.31551. Epub 2018 May 22. PMID 29786848
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Angelini DF, Ottone T, Guerrera G, Lavorgna S, Cittadini M, Buccisano F, De Bardi M, Gargano F, Maurillo L, Divona M, Noguera NI, Consalvo MI, Borsellino G, Bernardi G, Amadori S, Venditti A, Battistini L, Lo-Coco F. A Leukemia-Associated CD34/CD123/CD25/CD99+ Immunophenotype Identifies FLT3-Mutated Clones in Acute Myeloid Leukemia. Clin Cancer Res. 2015 Sep 1;21(17):3977-85. doi: 10.1158/1078-0432.CCR-14-3186. Epub 2015 May 8. PMID 25957287
- [Background] Yildirim E, Kirby JE, Brown DE, Mercier FE, Sadreyev RI, Scadden DT, Lee JT. Xist RNA is a potent suppressor of hematologic cancer in mice. Cell. 2013 Feb 14;152(4):727-42. doi: 10.1016/j.cell.2013.01.034. PMID 23415223
- [Background] Brown CJ, Hendrich BD, Rupert JL, Lafreniere RG, Xing Y, Lawrence J, Willard HF. The human XIST gene: analysis of a 17 kb inactive X-specific RNA that contains conserved repeats and is highly localized within the nucleus. Cell. 1992 Oct 30;71(3):527-42. doi: 10.1016/0092-8674(92)90520-m. PMID 1423611
- [Background] Wutz A, Rasmussen TP, Jaenisch R. Chromosomal silencing and localization are mediated by different domains of Xist RNA. Nat Genet. 2002 Feb;30(2):167-74. doi: 10.1038/ng820. Epub 2002 Jan 7. PMID 11780141
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254